CLINICAL TRIAL: NCT07318350
Title: Phase 3, Multicenter, Randomized, Parallel-group, Open-label, Non-inferiority Study of N0783 Versus Comparator (Formoterol 6 mcg / Budesonide 200 mcg) in the Treatment of Moderate Asthma
Brief Title: Study of Formoterol 6 mcg/Fluticasone 125 mcg by Eurofarma Laboratórios S.A. Versus Alenia® 6 mcg/200 mcg in Patients With Asthma (FORASMA)
Acronym: FORASMA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF195
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Moderate Asthma
Keywords: Asthma; Moderate Asthma; Alenia®; Non-inferiority; Randomized Clinical Trial; Phase 3
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N0783 (Experimental): Participants will receive N0783 administered via inhalation according to the dosing regimen specified in the protocol for the treatment of moderate asthma.
  Interventions: Drug: N0783
- Alenia® (Active Comparator): Participants will receive Alenia® (Formoterol 6 mcg / Budesonide 200 mcg) administered via inhalation according to the dosing regimen specified in the protocol for the treatment of moderate asthma.
  Interventions: Drug: Alenia® (Formoterol 6 mcg / Budesonide 200 mcg)

INTERVENTIONS:
Drug: N0783 — N0783 is a fixed-dose combination administered via inhalation using a metered-dose inhaler. Participants will receive the study drug according to the dosing regimen specified in the protocol for the treatment of moderate asthma.
  Arms: N0783
Drug: Alenia® (Formoterol 6 mcg / Budesonide 200 mcg) — Alenia® is a fixed-dose combination of Formoterol 6 mcg and Budesonide 200 mcg administered via inhalation using a metered-dose inhaler. Participants will receive the comparator drug according to the dosing regimen specified in the protocol for the treatment of moderate asthma.
  Arms: Alenia®

SUMMARY:
This is a Phase 3, multicenter, randomized, parallel-group, open-label, non-inferiority clinical trial designed to evaluate the efficacy and safety of N0783 compared to Alenia® (Formoterol 6 mcg / Budesonide 200 mcg) in the treatment of moderate asthma. Adult patients diagnosed with moderate asthma according to clinical and functional criteria will be enrolled. The primary objective is to demonstrate that N0783 is not inferior to Alenia® in improving asthma control. Participants will receive treatment according to the assigned intervention and will be monitored through scheduled visits for assessment of lung function, symptom control, and safety parameters throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and ≤ 65 years at Screening.
* History of recurrent asthma symptoms (cough, wheezing, shortness of breath, chest tightness).
* Previous medical diagnosis of asthma (confirmed by records, prescriptions, or participant report).
* Documented reversible airway obstruction by spirometry: FEV₁ increase ≥ 200 mL and ≥ 12% post-bronchodilator (at screening or prior report).
* Moderate asthma (GINA step 3) for ≥ 6 months, clinically stable and controlled with LABA + low-dose inhaled corticosteroid for ≥ 90 days.
* ACQ-7 score ≤ 0.75 at Screening.
* At Randomization: ACQ-7 score ≤ 0.75 and ≥ 70% adherence during run-in.

Exclusion Criteria:

* Moderate/severe asthma exacerbation within 90 days prior to screening.
* Other pulmonary disease (including predominant COPD).
* Symptomatic acute or chronic respiratory infection.
* BMI ≥ 40 kg/m².
* Use of LAMA within 6 months prior to screening.
* Oral or depot corticosteroids within 30 days prior to screening.
* Biologic therapy for asthma, allergic rhinitis, or urticaria within 12 months prior to screening.
* Systemic vasoconstrictors within 7 days prior to screening.
* Known hypersensitivity to formoterol, fluticasone, budesonide, or any component of study drugs.
* Active pulmonary tuberculosis or fungal airway infection.
* History or presence of ischemic heart disease, severe arrhythmias, cardiac decompensation, idiopathic subvalvular aortic stenosis, severe hypertension, aneurysm, pheochromocytoma, hypertrophic obstructive cardiomyopathy, thyrotoxicosis, QTc > 450 ms.
* History of hyperthyroidism or uncontrolled diabetes mellitus.
* Severe or uncontrolled disease at investigator's discretion.
* Pregnancy or breastfeeding; women of childbearing potential not using effective contraception.
* Participation in another clinical trial within 12 months unless direct benefit expected.
* Any condition making participant unsuitable for study per investigator.
* At Randomization: asthma exacerbation during run-in, prohibited medication use, HbA1c ≥ 10%, TSH below normal, ALT or AST > 2× ULN, serum potassium below normal, severe renal impairment (eGFR < 30 mL/min/1.73m²), clinically significant ECG changes or QTc > 450 ms, or any abnormality making participant unsuitable.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Absolute change in pre-bronchodilator FEV₁ (L) from baseline to Week 12 | 12 weeks after treatment initiation
  Improvement in pre-bronchodilator forced expiratory volume in one second (FEV₁), assessed by spirometry. The absolute change in FEV₁ (in liters) will be measured at Week 12 (Final Visit) compared to baseline (Randomization Visit).